CLINICAL TRIAL: NCT01405209
Title: Variaciones En El Elctrocardiograma Como Prediccion Del Desarrollo De Fibrilacion AURIC
Brief Title: Electrocardiogram Variations in the Prediction of Development of Atrial Fibrillation
Acronym: EKG
Status: Completed | Type: Observational
Sponsor: Hospital Italiano de Buenos Aires (Other)
Responsible Party: Principal Investigator, Diego Hernan Giunta, MD, MD, Hospital Italiano de Buenos Aires
Other Study IDs: 1713
Record Dates: First submitted 2011-07-28; First posted 2011-07-29 (Estimated); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Atrial Fibrillation
Keywords: EKG; AF; biosignals
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Atrial Fibrillation: Patients who develop atrial fibrillation
- Non Atrial FIbrillation: Patients without atrial fibrillation

SUMMARY:
Atrial fibrillation (AF) is the most common arrhythmia, affecting 1% of adults, with its prevalence increasing with age [1]. It is associated with increased morbidity and mortality.

Most patients who develop AF have architectural and anisotropic micro changes in the atrial myocardium. These cause heterogeneous and discontinuous changes in the patterns of impulse propagation, heterogeneous atrial activation and shortening of atrial refractory period [2, 3].

Since 1911 the standard EKG [4] (approximately 15 seconds of recording and bandwidth 0.05 to 150 Hz) is the most used tool for the evaluation of patients with arrhythmias, due to its low cost and high availability. Various electrocardiographic patterns are known predictors of AF as evidenced by direct visual inspection. For example, prolongation of P wave duration during sinus rhythm would correlate with structural changes such as increasing the size of the left atrium (the increase in left atrial pressure) or a decrease in driving time [5]. These changes favor the development of reentry circuits responsible for the development and maintenance of AF.

The registration of the electrocardiographic activity provides much more information than evidenced by direct visual inspection. Biosignal processing of these specific techniques to detect potential delays caused by abnormal conduction of the myocardium that favor re-entry mechanisms [6-10]. For this purpose prolonged ECG with 1000 Hz sampling frequency. Knowledge about the prediction of the development of AF with the standard ECG is not obvious on visual inspection is limited.

Many of these structural changes and anisotropic, occur slowly over time and may be evidenced by direct variations between 2 ECG from the same individual [11]. Little is known about whether differences in morphology, axis, scope or duration of P wave related to these structural changes may predict the development of AF.

Our main purpose is to evaluate the prognostic performance of a set of parameters as evidenced by direct inspection of the ECG, and ECG changes from 2 to predict the FA development. The design of this tool could allow future generation of software capable of identifying and reporting these variations, most useful prognostic risk in patients with AF.

DETAILED DESCRIPTION:
Retrospective cohort of patients 18 years or older with 2 EKG with sinusal rithm between 2004 - 2011.

ELIGIBILITY:
Inclusion Criteria:

1. Patients over 18 years Health Plan members of the Italian Hospital of Buenos Aires with at least 2 ECG separated .

Exclusion Criteria:

1. Patients with sinus rhythm different.
2. Patients with a history of congenital heart disease (tetralogy of fallot, CIA)
3. Patients with implanted defibrillator or pacemaker.
4. Patients with a history of cardiac surgery or performing heart surgery from the last ECG and the development of AF.
5. Patients with a history of radiofrequency ablation for treatment of arrhythmias.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients belonging to Health Plan Hospital Italiano de Buenos Aires active members who have ambulatory monitoring after the last follow-up ECG
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2011-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Variations (differences or deltas) between 2 standard ECG separated in time | at least 20 days after the first ekg
  To describe and evaluate the association between the variations (differences or deltas) between 2 standard ECG separated in time (eg difference in p-wave amplitude, difference in wavelength p) to predict development of AF

CONTACTS AND LOCATIONS:
Overall Officials: Diego H Giunta, MD, Principal Investigator — Hospital Italiano de Buenos Aires
Locations (1):
- Hospital Italiano de Buenos AIres, Buenos Aires, Argentina